CLINICAL TRIAL: NCT01116739
Title: Preventing Caries in Preschoolers: Testing a Unique Service Delivery Model in American Indian Head Start Programs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-0892; 1U54DE019259 (NIH)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Fluoride Varnish and Oral Health Promotion; Usual Care
MeSH Terms: interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COHS administered fluoride varnish and oral health education (Experimental): Paraprofessionals, called community oral health specialists (COHS), will be trained to administer fluoride varnish and oral health education to head start children quarterly for 2 years.
  Interventions: Device: Fluoride varnish; Behavioral: Oral health education
- Usual care (Active Comparator): Usual care will include regular dental services provided by the Indian Health Service.
  Interventions: Other: Dental services delivered by the Indian Health Service.

INTERVENTIONS:
Device: Fluoride varnish — Fluoride varnish will be administered by the COHS quarterly for 2 years.
  Arms: COHS administered fluoride varnish and oral health education
Behavioral: Oral health education — Oral health education will be provided quarterly for 2 years. It will include information about how to mitigate the known risk factors for early childhood dental caries.
  Arms: COHS administered fluoride varnish and oral health education
Other: Dental services delivered by the Indian Health Service.
  Arms: Usual care

SUMMARY:
An intensive intervention of specially trained paraprofessionals, called community oral health specialists (COHS), administering on a quarterly basis for 2 years fluoride varnish and oral health promotion education, compared to usual care, will reduce decayed, missing, and filled tooth surface measures at 2 years for children in American Indian Head Start Programs.

DETAILED DESCRIPTION:
The study design will be a clustered randomized design. Fifty-two head start classes in a Southwest American Indian Reservation will be randomized, 26 to the intervention program and 26 to usual care. The intervention will be comprised of specially trained paraprofessionals, called community oral health specialists (COHS), administering fluoride varnish and oral health promotion education quarterly for 2 years. Baseline and annual measures of decayed, missing, and filled tooth surfaces (dmfs) of the children, and surveys of their caregivers' dental knowledge, attitudes, and behaviors will be completed. The study will be a 5-year study, with 2 years for intake/accrual, and 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-5 enrolled in Head Start Centers on a Southwest Indian Reservation and having a primary caregiver (preferably mother, or the child's legal guardian as documented by the HSC)
* American Indian, as defined by the tribe, or
* Children of other racial/ethnic groups who are in the Head Start classes on the Reservation
* Parent/caregiver able to read, understand, and sign the study consent form, and
* Willing and able to follow the study procedures and instructions

Exclusion Criteria:

* Allergy to any of the components of the fluoride varnish
* Ulcerative gingivitis
* Stomatitis
* Other conditions resulting in disrupted or irritated oral mucosa
* Any other conditions or findings that, in the opinion of the investigators, would interfere with or preclude participation in the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2060 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Braun, MD MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Background] Quissell DO, Bryant LL, Braun PA, Cudeii D, Johs N, Smith VL, George C, Henderson WG, Albino J. Preventing caries in preschoolers: successful initiation of an innovative community-based clinical trial in Navajo Nation Head Start. Contemp Clin Trials. 2014 Mar;37(2):242-51. doi: 10.1016/j.cct.2014.01.004. Epub 2014 Jan 25. PMID 24469238
- [Result] Albino J, Tiwari T, Henderson WG, Thomas J, Bryant LL, Batliner TS, Braun PA, Wilson A, Quissell DO. Learning from caries-free children in a high-caries American Indian population. J Public Health Dent. 2014 Fall;74(4):293-300. doi: 10.1111/jphd.12058. Epub 2014 Jun 24. PMID 24961881
- [Result] Batliner T, Wilson AR, Tiwari T, Glueck D, Henderson W, Thomas J, Braun P, Cudeii D, Quissell D, Albino J. Oral health status in Navajo Nation Head Start children. J Public Health Dent. 2014 Fall;74(4):317-25. doi: 10.1111/jphd.12061. Epub 2014 Jun 23. PMID 24954053
- [Result] Braun PA, Lind KE, Henderson WG, Brega AG, Quissell DO, Albino J. Validation of a pediatric oral health-related quality of life scale in Navajo children. Qual Life Res. 2015 Jan;24(1):231-9. doi: 10.1007/s11136-014-0751-3. Epub 2014 Jul 9. PMID 25005885
- [Result] Tiwari T, Casciello A, Gansky SA, Henshaw M, Ramos-Gomez F, Rasmussen M, Garcia RI, Albino J, Batliner TS; Early Childhood Caries Collaborating Centers. Recruitment for health disparities preventive intervention trials: the early childhood caries collaborating centers. Prev Chronic Dis. 2014 Aug 7;11:E133. doi: 10.5888/pcd11.140140. PMID 25101490
- [Result] Tiwari T, Quissell DO, Henderson WG, Thomas JF, Bryant LL, Braun PA, Albino JE. Factors Associated with Oral Health Status in American Indian Children. J Racial Ethn Health Disparities. 2014 Sep 1;1(3):148-156. doi: 10.1007/s40615-014-0017-3. PMID 25232515
- [Result] Braun PA, Quissell DO, Henderson WG, Bryant LL, Gregorich SE, George C, Toledo N, Cudeii D, Smith V, Johs N, Cheng J, Rasmussen M, Cheng NF, Santo W, Batliner T, Wilson A, Brega A, Roan R, Lind K, Tiwari T, Shain S, Schaffer G, Harper M, Manson SM, Albino J. A Cluster-Randomized, Community-Based, Tribally Delivered Oral Health Promotion Trial in Navajo Head Start Children. J Dent Res. 2016 Oct;95(11):1237-44. doi: 10.1177/0022034516658612. Epub 2016 Jul 20. PMID 27439724
- [Derived] Wilson AR, Tiwari T, Thomas JF, Henderson WG, Braun PA, Albino J. Validation of Psychosocial Measures Assessing American Indian Parental Beliefs Related to Control over Their Children's Oral Health. Int J Environ Res Public Health. 2020 Jan 8;17(2):403. doi: 10.3390/ijerph17020403. PMID 31936256
- [Derived] Albino J, Tiwari T, Gansky SA, Henshaw MM, Barker JC, Brega AG, Gregorich SE, Heaton B, Batliner TS, Borrelli B, Geltman P, Kressin NR, Weintraub JA, Finlayson TL, Garcia RI; Early Childhood Caries Collaborating Centers. The basic research factors questionnaire for studying early childhood caries. BMC Oral Health. 2017 May 19;17(1):83. doi: 10.1186/s12903-017-0374-5. PMID 28526003

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care will include regular dental services provided by the Indian Health Service.
  Dental services delivered by the Indian Health Service.
Period: Overall Study
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Started | 1056 | 1004
Completed | 926 | 868
Not Completed | 130 | 136
Not completed — Child had 2 years of HS | 110 | 128
Not completed — Withdrawal by Subject | 6 | 0
Not completed — child too young | 2 | 6
Not completed — child not enrolled in head start | 10 | 2
Not completed — enrolled caregiver not legal guardian | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics data was collected for participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care | Total
Number analyzed (Participants) | 926 | 868 | 1794
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 463 | 434 | 897
  Between 18 and 65 years | 463 | 434 | 897
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 621 | 582 | 1203
  Male | 305 | 286 | 591
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 926 | 868 | 1794
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 926 | 868 | 1794
Child Enrolled in a Head Start program in one of 53 centers on the Navajo Nation [Count of Participants; unit: Participants] | 926 | 868 | 1794

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Decayed, Missing, and Filled Tooth Surfaces (Dmfs) at Baseline
Description: The number of decayed, missing, and filled tooth surfaces (dmfs) for each child. The dental examiners will be trained and calibrated, and standardized criteria and instruments will be used for the detection of the dental caries.
Time Frame: Baseline
Population: Only children, not parents, were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: dmfs
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 443 | 424
dmfs | 19.9 (20.1) | 22.8 (20.1)

2. Primary Outcome: Evaluation of Decayed, Missing, and Filled Tooth Surfaces (Dmfs) at Year 1
Description: as for outcome 1
Time Frame: 1 Year
Population: Only children, not parents, were analyzed for this outcome measure. Some participants were unavailable for analysis at this timepoint.
Measure: Mean (Standard Deviation); unit: dmfs
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 217 | 231
dmfs | 23.3 (20.4) | 27.1 (21.5)

3. Primary Outcome: Evaluation of Decayed, Missing, and Filled Tooth Surfaces (Dmfs) at Year 2
Description: as for outcome 1
Time Frame: 2 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dmfs
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 238 | 229
dmfs | 28.5 (21.1) | 31.2 (21.3)

4. Primary Outcome: Evaluation of Decayed, Missing, and Filled Tooth Surfaces (Dmfs) at Year 3
Description: as for outcome 1
Time Frame: 3 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dmfs
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 118 | 111
dmfs | 32.8 (22.3) | 33.6 (18.6)

5. Secondary Outcome: Acquisition of Dental Attitudes and Behaviors of the Caregivers of the Children
Description: An automated computer assisted survey interview (ACASI)will be done of the caregivers of the children. The questions have been standardized across 6 studies from the Collaborating Research Centers to Reduce Oral Health Disparities. The survey assessing attitudes and behaviors is comprised of 12 items. Scores are calculated as a percentage of appropriate responses. Therefore, possible scores range from 0-100.
Time Frame: Over 3 years
Population: Only the caregivers, not the children, were analyzed for this outcome measure. Not all participants were available for analysis at every time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 463 | 434
score on a scale
  Baseline | 54.4 (19.3) | 56.1 (18.3)
  Year 1: number analyzed (Participants) | 221 | 230
  Year 1 | 62.7 (18.8) | 58.2 (19.6)
  Year 2: number analyzed (Participants) | 233 | 225
  Year 2 | 63.4 (18.7) | 61.1 (18.3)
  Year 3: number analyzed (Participants) | 110 | 115
  Year 3 | 65.6 (18.9) | 66.4 (17.6)

6. Secondary Outcome: Evaluation of Caries Patterns
Description: Caries patterns will be studied in terms of the specific teeth and tooth surfaces that are affected. Caries prevalence is defined as the presence of more than 0 dmfs (decayed, missing, or filled surfaces) in the child participant. The percentage of child participants with caries prevalence is reported.
Time Frame: Over 3 years
Population: Only children, not parents, were analyzed for this outcome measure. Some participants were unavailable for analysis at each timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 443 | 424
percentage of participants
  Baseline | 86.5 | 90.1
  Year 1: number analyzed (Participants) | 217 | 231
  Year 1 | 89.9 | 90.9
  Year 2: number analyzed (Participants) | 238 | 229
  Year 2 | 95.4 | 96.1
  Year 3: number analyzed (Participants) | 118 | 111
  Year 3 | 96.6 | 98.2

7. Secondary Outcome: Comparison of Utilization and Costs of Dental Care
Description: Utilization and costs of dental care received by the children in the study will be compared, as well as the costs of the intervention program.
Time Frame: Up to 3 years after randomization
Population: Cost and utilization outcome measure data was not collected.
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Acquisition of Dental Knowledge of the Caregivers of the Children
Description: An automated computer assisted survey interview (ACASI)will be done of the caregivers of the children. The questions have been standardized across 6 studies from the Collaborating Research Centers to Reduce Oral Health Disparities. The survey assessing knowledge is comprised of 14 items. Scores are calculated as a percentage of correct answers. Therefore, possible scores range from 0-100.
Time Frame: Over 3 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
Number analyzed (Participants) | 463 | 434
score on a scale
  Baseline | 75.1 (30.7) | 73.6 (13.1)
  Year 1: number analyzed (Participants) | 221 | 230
  Year 1 | 80.4 (13.1) | 76.8 (13.5)
  Year 2: number analyzed (Participants) | 233 | 225
  Year 2 | 81.4 (14.8) | 78.0 (13.2)
  Year 3: number analyzed (Participants) | 110 | 115
  Year 3 | 81.2 (13.4) | 79.5 (12.8)

ADVERSE EVENTS:
Time Frame: 3 Years
Arm/Group | COHS Administered Fluoride Varnish and Oral Health Education | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/926 | 0/868
Serious Adverse Events (participants affected / at risk) | 0/926 | 0/868
Other Adverse Events (participants affected / at risk) | 0/926 | 0/868

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT01116739/Prot_SAP_000.pdf